CLINICAL TRIAL: NCT00402077
Title: A Randomized, Parallel-Group, Multicenter Study to Examine the Safety, Tolerability, and Body Weight Effect of Subcutaneous Pramlintide Alone and in Combination With the Oral Antiobesity Agents Sibutramine or Phentermine in Overweight and Obese Subjects
Brief Title: A Study to Examine the Safety, Tolerability, and Body Weight Effect of Pramlintide Alone and in Combination With Oral Antiobesity Agents in Overweight and Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFA203
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; pramlintide; Symlin; sibutramine; Meridia; phentermine; Amylin
MeSH Terms: conditions — Overweight; Obesity | interventions — pramlintide; sibutramine; Phentermine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: pramlintide acetate
- 2 (Experimental)
  Interventions: Drug: pramlintide acetate; Drug: sibutramine
- 3 (Experimental)
  Interventions: Drug: pramlintide acetate; Drug: phentermine
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pramlintide acetate — subcutaneous injection, three times a day, 120mcg
  Other Names: Symlin
  Arms: 1; 2; 3
Drug: sibutramine — oral tablet, once a day, 10mg
  Other Names: Meridia
  Arms: 2
Drug: phentermine — oral tablet, once a day, 37.5mg
  Other Names: Adipex-P; Fastin; Obenix; Oby-Trim
  Arms: 3
Drug: placebo — subcutaneous injection, three times a day
  Arms: 4

SUMMARY:
This study will examine the safety, tolerability, and body weight effect of subcutaneous pramlintide alone and in various combinations with the oral antiobesity agents sibutramine or phentermine in overweight and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Is obese with a Body Mass Index (BMI) >=30 kg/m^2 to <=50 kg/m^2 or overweight with a BMI >=27 kg/m^2 in the presence of other risk factors (e.g., hyperlipidemia, sleep apnea, or treatment for these conditions)
* Has been obese or overweight for at least one year prior to study start
* Either is not treated with or has been on a stable treatment regimen with any of the following medications for a minimum of 2 months prior to study start: *hormone replacement therapy; *oral contraceptives; *lipid-lowering agents; *thyroid replacement therapy; *metformin

Exclusion Criteria:

* Is currently enrolled in or is planning to enroll in a formal weight-loss program
* Is unwilling or unable to participate in a lifestyle intervention program as part of the study
* Has been treated (within the 2 months prior to study start), is currently treated, or is expected to require or undergo treatment with any of the following excluded medications: *prescription or over the counter antiobesity agents (within the 6 months prior to study start); *psychotropic/neurological agents (i.e., antipsychotic, antiepileptic, antidepressant, or antianxiety agents, or mood stabilizers); *steroids that are known to result in high systemic absorption; *calcitonin; *ketoconazole; *antidiabetic medications
* Has had liposuction, abdominoplasty, or a similar procedure within 1 year before study start or is planning to have such a procedure during the study
* Has received any investigational drug within 1 month (or 5 half-lives of investigational drug, whichever is greater) before study start
* Has previously used pramlintide either by prescription or as part of a clinical study
* Has used sibutramine or phentermine (either by prescription or as part of a clinical study) within 2 years before study start
* Has donated blood within 2 months before study start, or is planning to donate blood during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
All treatment-emergent adverse events occurring during the 24-week treatment period | 24 weeks
Absolute change in body weight from baseline to Week 12 | 12 weeks

SECONDARY OUTCOMES:
Percent change in body weight from baseline to Week 12 | 12 weeks
Percentage of subjects achieving at least 5% weight loss from baseline to Week 12 and Week 24 | 24 weeks
Absolute and percent changes in body weight from baseline to Week 2, Week 4, Week 8, Week 16, Week 20, and Week 24 | 24 weeks
Absolute changes in anthropometric measurements (hip and waist circumferences) from baseline to Week 12 and Week 24 | 24 weeks
Changes in fasting serum concentrations of lipids from baseline to Week 12 and Week 24 | 24 weeks
Changes in summary measures derived from patient reported outcome questionnaires from baseline to Week 12 and Week 24 | 24 weeks
Changes in individual item responses from patient reported outcome questionnaires from baseline to Week 12 and Week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (16):
- United States (16):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Chula Vista, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Walnut Creek, California
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Louisville, Kentucky
  - Research Site, New York, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Eugene, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas